CLINICAL TRIAL: NCT05022186
Title: Comparative Randomized Clinical Trial of the Efficacy of Cannabidiol and Homotaurine in Patients With Mild Cognitive Impairment and APOE ε4 Carriers
Brief Title: The Effects of Cannabidiol and Homotaurine in Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek Alzheimer's Association and Related Disorders (Other)
Responsible Party: Principal Investigator, Magda Tsolaki, Professor of Neurology, Medical School, Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 65/06-02-2021
Record Dates: First submitted 2021-04-27; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment
Keywords: cannabidiol; homotaurine; Mild Cognitive Impairment; Cognition; Mental Health
MeSH Terms: conditions — Cognitive Dysfunction; Psychological Well-Being | interventions — Cannabidiol; 5''-hydroxycannabidiol glucoside; tramiprosate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group receiving Cannabidiol (Experimental): These patients will receive cannabidiol 5% without other medication for cognition and depression
  Interventions: Drug: Cannabidiol Oil
- Group receiving Homotaurine (Experimental): These patients will receive Vivimind (homotaurine) without other medication for memory and depression
  Interventions: Drug: Homotaurine
- Control group (No Intervention): These patients will not receive treatment

INTERVENTIONS:
Drug: Cannabidiol Oil — Patients will use it with specific instructions and they will be monitored at least one time in a month
  Other Names: CBD 5%
  Arms: Group receiving Cannabidiol
Drug: Homotaurine — Patients will use it with specific instructions and they will be monitored at least one time in a month
  Other Names: Vivimind
  Arms: Group receiving Homotaurine

SUMMARY:
A Randomized Clinical Trial that will compare the effects of Cannabidiol and Homotaurine in cognition and mental health in patients with Mild Cognitive Impairment and APOE ε4 carriers. Ninety patients will be recruited and they will be randomly distributed in three groups. The first group will receive treatment with Cannabidiol 5%, the second group will receive treatment with Vivimind and the third group will not receive any treatment. The three groups will be compared by using an extensive neuropsychological examination and biomarkers' results from cerebrospinal fluid and blood

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment
* Carry APOE ε4 gene

Exclusion Criteria:

* Diagnosis of Dementia
* Patients who receive medication for memory or depression
* Patients who do not carry APOE ε4 gene

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Mini Mental State Examination (MMSE) score | 12-24 months
Changes in Montreal Cognitive Assessment (MoCA) score | 12-24 months
  Screening test to assess general cognitive function
Changes in Functional Cognitive Assessment (FUCAS) score | 12-24 months
  Measurement of daily functionality
Changes in Letter & Category Verbal Fluency | 12-24 months
  Measurement of verbal fluency, learning, long term memory and categorization skills
Changes in Clinical Dementia Rating Scale score | 12-24 months
  Measurement of general cognitive function
Changes in ADAS-COG | 12-24 months
  Measurement of general cognitive function
Changes in Rey Auditory Verbal Learning Test | 12-24 months
  Screening tool to assess verbal memory and learning
Changes in Rey Osterrieth Complex Figure | 12-24 months
  Screening tool to assess visuospatial memory
Changes in Functional Rating Scale for Dementia | 12-24 months
  Measurement of daily functionality
Changes in Trail Making Test A & B | 12-24 months
  Screening tool to assess working memory and processing speed
Changes in Geriatric Depression Scale | 12-24 months
  Screening tool to assess depressive symptoms
Changes in SAST | 12-24 months
  Screening tool to assess anxiety
Changes in Beck Anxiety Inventory | 12-24 months
  Screening tool to assess anxiety
Changes in Rivermead Behavioural Memory Test | 12-24 months
  Screening tool to assess episodic memory and learning
Changes in STROOP Test | 12-24 months
  Measurement of selective attention and cognitive flexibility
Changes in Symbol-Digit Test | 12-24 months
  Measurement of processing speed, learning and working memory
Changes in BDNF | 12-24 months
  Cerebrospinal Fluid Biomarker
Changes in MDA | 12-24 months
  Cerebrospinal Fluid Biomarker
Changes in GFAP | 12-24 months
  Cerebrospinal Fluid Biomarker
Changes in Tau-protein | 12-24 months
  Cerebrospinal Fluid Biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Greek Association of Alzheimer's Disease and Related Disorders, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Participants' personal data will not be shared with other researchers